CLINICAL TRIAL: NCT03729687
Title: Phase II of Short Course Radiation Therapy Followed by Pre-operative Chemotherapy and Surgery in Primary High-risk Rectal Cancer
Brief Title: Short Course Radiation Therapy Followed by Pre-operative Chemotherapy and Surgery in High-risk Rectal Cancer
Acronym: LARCT-US
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Collaborators: Swedish Cancer Society (Other)
Responsible Party: Principal Investigator, Bengt Glimelius, Senior Professor, consultant, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LARCT-US v1.3
Record Dates: First submitted 2018-10-10; First posted 2018-11-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; high risk; total neoadjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Treatment with short-course radiotherapy (scRT) followed by 4 cycles of CAPOX chemotherapy and surgery in locally advanced rectal cancer while waiting for the results of the randomized phase III RAPIDO trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LARCT-US (Experimental): Short Course Radiation Therapy (5 x 5 Gy in 1 week, scRT) followed by 4 cycles of Pre-operative Chemotherapy using capecitabine and oxaliplatin (CAPOX) and Surgery in High-risk Rectal Cancer
  Interventions: Combination Product: radiotherapy, capecitabine, oxaliplatin

INTERVENTIONS:
Combination Product: radiotherapy, capecitabine, oxaliplatin — 5x5 Gy radiotherapy in 1 week, 4 cycles of CAPOX (capecitabine 1000 mg/m2 x2 d 1-14, oxaliplatin 130 mg/m2 d 1 every third week), surgery

SUMMARY:
Patients with a primary rectal cancer without detectable distant metastasis who after locoregional therapy only, meaning preoperative radio(chemo)therapy plus surgery have at least a 40% risk of not having a CRM negative resection or a recurrence, local or distant, within three years will be treated with the short course 5 x 5 Gy radiation scheme followed by four cycles of combination chemotherapy (capecitabine and oxaliplatin) and TME surgery

DETAILED DESCRIPTION:
The multicentre, multinational RAPIDO (Rectal cancer And Pre-operative Induction therapy followed by Dedicated Operation, EudraCT number 2010-023957-12) closed patient entry in June 2016 after having randomised the planned number of 920 patients. In the study, patients were randomised to conventional chemoradiotherapy (CRT) to 50 Gy with capecitabine followed by surgery or to short-course radiotherapy (scRT, 5 x 5 Gy), 6 cycles of oxaliplatin-capecitabine (CAPOX) followed by surgery. In the CRT arm, adjuvant chemotherapy with 8 cycles of CAPOX was optional. At the time of closure of the RAPIDO study, it was discussed in Uppsala whether CRT should be the reference treatment for these high-risk rectal cancers, the experimental treatment or an alternative. Influenced by a Polish study reported by Bujko et al in 2016 with a similar design comparing CRT with scRT followed by 3 cycles of FOLFOX), it was decided that the reference treatment for patient with primary rectal cancer at high risk of failing either locally or systemically should be scRT followed by 4 cycles of CAPOX and surgery. This regimen, identical to the experimental arm in a Chinese trial (Stellar trial (ClinicalTrials.gov NCT02533271), preliminarily revealing promising pCR rates has since then been the reference treatment for patients having the same inclusion criteria as in the RAPIDO trial. Other centres in Sweden have also decided to use this regimen as reference treatment. A formal protocol is written and approved.

ELIGIBILITY:
Inclusion Criteria:

* • Histological proof of newly diagnosed primary adenocarcinoma of the rectum

  * Locally advanced tumour fulfilling at least one of the following criteria on pelvic MRI indicating high risk of failing locally and/or systemically (T4b, i.e. overgrowth to an adjacent organ or structure like the prostate, urinary bladder, uterus, sacrum, pelvic floor or side-wall (according to TNM version 7), cT4a, i.e. peritoneal involvement, extramural vascular invasion (EMVI+). N2, i.e. four or more lymph nodes in the mesorectum showing morphological signs on MRI indicating metastatic disease. Four or more nodes, whether enlarged or not, with a rounded, homogeneous appearance is thus not sufficient. Positive MRF, i.e. tumour or lymph node < 1 mm from the mesorectal fascia. Enlarged lateral nodes, > 1 cm (lat LN+).

Exclusion Criteria:

* Extensive growth into cranial part of the sacrum (above S3) or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumour down-sizing is seen.
* Presence of metastatic disease or recurrent rectal tumour. Familial Adenomatosis Polyposis coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative Colitis.
* Concomitant malignancies, except for adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri. Subjects with prior malignancies must be disease-free for at least 5 years.
* Known DPD deficiency.
* Any contraindications to MRI (e.g. patients with pacemakers).
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Concurrent uncontrolled medical conditions.
* Any investigational treatment for rectal cancer within the past month.
* Pregnancy or breast feeding.
* Patients with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac dysrhythmia, e.g. atrial fibrillation, even if controlled with medication) or myocardial infarction within the past 12 months.
* Patients with symptoms of peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate and clinical complete response (cCR) rate | pCR assessed directly after surgery and cCR 12 months after end of treatment if no surgery is performed (cCR)]
  pCR assessed at pathological examination of the surgical specimen, cCR at clinical and radiological (MRI) examination

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  non-radical surgery, recurrence or death within 3 years
Neoadjuvant rectal score (NAR score) | After surgery when the patological examination of the surgical specimen is completed
  Score from 0 - 100, where 0 is best
Incidence of Treatment-Emergent Adverse Events | within 60 days after end of treatment
  CTCAE v 4.0
Long-term Adverse Events | 4 years after end of treatment
  CTCAE v 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Glimelius, MD,PhD, Principal Investigator — Uppsala University
Locations (1):
- Akademiska sjukhuset, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson PJ, van Etten B, Hospers GA, Pahlman L, van de Velde CJ, Beets-Tan RG, Blomqvist L, Beukema JC, Kapiteijn E, Marijnen CA, Nagtegaal ID, Wiggers T, Glimelius B. Short-course radiotherapy followed by neo-adjuvant chemotherapy in locally advanced rectal cancer--the RAPIDO trial. BMC Cancer. 2013 Jun 7;13:279. doi: 10.1186/1471-2407-13-279. PMID 23742033
- [Background] Bujko K, Wyrwicz L, Rutkowski A, Malinowska M, Pietrzak L, Krynski J, Michalski W, Oledzki J, Kusnierz J, Zajac L, Bednarczyk M, Szczepkowski M, Tarnowski W, Kosakowska E, Zwolinski J, Winiarek M, Wisniowska K, Partycki M, Beczkowska K, Polkowski W, Stylinski R, Wierzbicki R, Bury P, Jankiewicz M, Paprota K, Lewicka M, Cisel B, Skorzewska M, Mielko J, Bebenek M, Maciejczyk A, Kapturkiewicz B, Dybko A, Hajac L, Wojnar A, Lesniak T, Zygulska J, Jantner D, Chudyba E, Zegarski W, Las-Jankowska M, Jankowski M, Kolodziejski L, Radkowski A, Zelazowska-Omiotek U, Czeremszynska B, Kepka L, Kolb-Sielecki J, Toczko Z, Fedorowicz Z, Dziki A, Danek A, Nawrocki G, Sopylo R, Markiewicz W, Kedzierawski P, Wydmanski J; Polish Colorectal Study Group. Long-course oxaliplatin-based preoperative chemoradiation versus 5 x 5 Gy and consolidation chemotherapy for cT4 or fixed cT3 rectal cancer: results of a randomized phase III study. Ann Oncol. 2016 May;27(5):834-42. doi: 10.1093/annonc/mdw062. Epub 2016 Feb 15. PMID 26884592

DOCUMENTS (1):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03729687/Prot_000.pdf